CLINICAL TRIAL: NCT01148823
Title: Influence of Time of Permanence of Dressing Following Breast Reconstruction on Skin Colonization and on Surgical Site Infection Rates
Brief Title: Time of Permanence of Dressing Following Breast Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daniela Francescato Veiga (Other)
Collaborators: Universidade do Vale do Sapucai (Other)
Responsible Party: Sponsor-Investigator, Daniela Francescato Veiga, Professor, Federal University of São Paulo
Organization: Federal University of São Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Micro01
Record Dates: First submitted 2010-06-21; First posted 2010-06-22 (Estimated); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Surgical Site Infection
Keywords: breast; plastic surgery; bandages; surgical site infection; skin colonization
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Postoperative day 1 (Experimental): Dressing was removed on the first postoperative day
  Interventions: Other: Incisions covered for 1 day
- Postoperative day 6 (Experimental): Dressing was removed on the 6th postoperative day
  Interventions: Other: Incisions covered for 6 days

INTERVENTIONS:
Other: Incisions covered for 1 day — Dressing was removed on the first postoperative day.
  Other Names: PO1
  Arms: Postoperative day 1
Other: Incisions covered for 6 days — Dressing was removed on the 6th postoperative day.
  Other Names: PO6
  Arms: Postoperative day 6

SUMMARY:
This randomized clinical trial was designed to assess the influence of time of dressing after breast reconstruction procedures on surgical site infections rates and skin colonization.

DETAILED DESCRIPTION:
The rates of surgical site infections (SSI) after clean operations range from 1 to 2%. However, infection rates in the breast surgical literature tend to be higher, with reported rates ranging from 2 to 30%. In plastic surgery operations, to minimize the risk of SSI is imperative, since even minor infections are able to complicate the healing process and harm the cosmetic result.

The Centers for Disease Control and Prevention has established guidelines for postoperative incision care. However, there is no recommendation to cover an incision closed primarily beyond 48 hours, nor on the appropriate time to shower or bathe with an uncovered incision. This remains an unresolved issue.

ELIGIBILITY:
Inclusion Criteria:

•candidate to immediate or delayed breast reconstruction after mastectomy or segmental mastectomy

Exclusion Criteria:

* use of antibiotics at the time of the operation
* presence of skin lesions on the surgical site
* body mass index over 35Kg/m2
* hard smoking

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2007-06 (Actual); Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Surgical site infection (SSI) | 30th postoperative day and one year after operation
  Patients are followed weekly by a masked surgeon in regard to SSI, until the 30th postoperative day.CDC's criteria and classification was adopted.Patients are reevaluated at the end of the first year after operation.

SECONDARY OUTCOMES:
Skin colonization | 6 days postoperatively
  Samples are collected to cultures before dressing (control) and at the 6th postoperative day
Patients self assessments | 2 weeks postoperatively
  Patients scored dressing wear time with regard to safety, comfort and convenience.

CONTACTS AND LOCATIONS:
Overall Officials: Daniela F Veiga, MD, PhD, Study Chair — Universidade do Vale do Sapucaí and Universidade Federal de São Paulo
Locations (1):
- Hospital das Clinicas Samuel Libânio, Universidade do Vale do Sapucaí, Pouso Alegre, Minas Gerais, Brazil

REFERENCES:
- [Background] Veiga DF, Veiga-Filho J, Damasceno CA, Sales EM, Morais TB, Almeida WE, Novo NF, Ferreira LM. Dressing wear time after breast reconstruction: study protocol for a randomized controlled trial. Trials. 2013 Feb 22;14:58. doi: 10.1186/1745-6215-14-58. PMID 23432779
- [Result] Veiga DF, Veiga-Filho J, Mendes DA, Sales AM, Damasceno Ca, Ferreira LM. Dressing wear time after breast reconstruction: preliminary results of a randomized controlled trial. Plastic and Reconstructive Surgery 131(5S): 119, 2013.
- [Result] Veiga DF, Damasceno CA, Veiga-Filho J, Paiva LF, Fonseca FE, Cabral IV, Pinto NL, Juliano Y, Ferreira LM. Dressing Wear Time after Breast Reconstruction: A Randomized Clinical Trial. PLoS One. 2016 Dec 2;11(12):e0166356. doi: 10.1371/journal.pone.0166356. eCollection 2016. PMID 27911904
- See also: Study Protocol — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC4148541/pdf/13063_2014_Article_2203.pdf